CLINICAL TRIAL: NCT05416775
Title: An Open-label, Multicenter Phase Ib/II Clinical Study of SHR-8068 Combined With Adebrelimab and Platinum-based Chemotherapy in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Phase Ib/II Study of SHR-8068 Injection in the Treatment of Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-II-201-NSCLC
Record Dates: First submitted 2022-05-27; First posted 2022-06-13 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-05

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Platinum Compounds

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, dose-finding and efficacy-expansion phase Ib/II study. The first stage is for dose finding, using modified 3+3 design; the second stage is for dose confirmation and efficacy expansion through randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-8068 in combination with adebrelimab (Experimental)
  Interventions: Drug: SHR-8068；Adebrelimab
- SHR-8068 in combination with adebrelimab and platinum-based chemotherapy (Experimental)
  Interventions: Drug: SHR-8068；adebrelimab and platinum-based chemotherapy
- Adebrelimab in combination with platinum-based chemotherapy (Experimental)
  Interventions: Drug: Adebrelimab；platinum-based chemotherapy

INTERVENTIONS:
Drug: SHR-8068；Adebrelimab — SHR-8068: Sterile Injection, 50mg/10mL, Intravenous Infusion Adebrelimab: injection, 600mg/12mL, intravenous infusion
  Arms: SHR-8068 in combination with adebrelimab
Drug: SHR-8068；adebrelimab and platinum-based chemotherapy — SHR-8068: Intravenous Infusion Adebrelimab: injection, intravenous infusion Pemetrexed disodium for injection: , intravenous drip Paclitaxel for injection (albumin-bound): intravenous drip Paclitaxel injection: intravenous drip Carboplatin injection: intravenous drip Cisplatin injection: intravenous drip
  Arms: SHR-8068 in combination with adebrelimab and platinum-based chemotherapy
Drug: Adebrelimab；platinum-based chemotherapy — Adebrelimab: intravenous infusion Pemetrexed disodium for injection: intravenous drip Paclitaxel for injection (albumin-bound): intravenous drip Paclitaxel injection: intravenous drip Carboplatin injection: intravenous drip Cisplatin injection: intravenous drip
  Arms: Adebrelimab in combination with platinum-based chemotherapy

SUMMARY:
To evaluate the tolerability and safety of SHR-8068 in combination with adebrelimab in subjects with advanced NSCLC To evaluate the efficacy of SHR-8068 in combination with adebrelimab and platinum-based chemotherapy in subjects with advanced NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old, both male and female
2. Stage 1: pathologically diagnosed, incurable NSCLC subjects who have failed standard treatment
3. Stage 2: have a histologically or cytologically confirmed diagnosis of relapsed or metastatic NSCLC; have not received prior systemic treatment for their recurrent or metastatic NSCLC; PD-L1 TPS <50% as confirmed by central laboratory
4. At least one measurable lesion based on RECIST v1.1 criteria
5. ECOG PS score: 0-1 points
6. Expected survival period ≥ 3 months
7. Good levels of organ function
8. Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

1. Patients with EGFR activating mutation, positive ALK fusion gene or known ROS1 fusion gene
2. Untreated brain metastases; or associated with meningeal metastases, spinal cord compression, etc.
3. Uncontrolled pleural, pericardial, or ascites with clinical symptoms
4. Severe bone damage caused by tumor bone metastasis
5. Suffering from other malignant tumors in the past 3 years or at the same time
6. Presence of any active or known autoimmune disease
7. Systemic treatment with corticosteroids or other immunosuppressants within 2 weeks before the first dose
8. Have clinical symptoms or diseases of the heart that are not well controlled
9. Serious infection occurred within 1 month before the first dose
10. Past or current active interstitial lung disease requiring treatment, non-infectious pneumonia requiring glucocorticoid system treatment; current active pneumonia or pulmonary function test confirmed severe impairment of pulmonary function
11. With active pulmonary tuberculosis
12. Known positive history of human immunodeficiency virus test or acquired immunodeficiency syndrome, known active viral hepatitis
13. Known history of inflammatory bowel disease
14. Inoculated with live attenuated vaccine within 28 days before the first dose
15. Known allergic reaction to other monoclonal antibodies
16. Received >30 Gy of pulmonary radiotherapy within 6 months before the first dose; received major surgical treatment, systemic chemotherapy, immunotherapy or other clinical trial drugs within 4 weeks before the first dose; within 2 weeks before the first dose Received palliative radiotherapy; oral molecularly targeted drugs, discontinued to less than 5 half-lives before first dose; failure to recover from toxicity and/or complications of previous interventions to NCI-CTC AE ≤1 degree
17. According to the judgment of the researcher, there are other factors that may affect the results of the study or cause the study to be terminated halfway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | The observation period is 21 days after the first dose
Objective Response Rate, determined using RECIST v1.1 criteria, defined as best overall response (complete or partial response) across all assessment time points; | up to 2 years

SECONDARY OUTCOMES:
Disease Control Rate, determined using RECIST v1.1 criteria | up to 2 years
Progression-Free-Survival assessed by investigator | up to 2 years

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Anhui Chest Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - West China Hospital Of Sichuan University, Chengdu, Chengdu
  - Cancer Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Affiliated Tumor Hospital of Shandong First Medical University, Jinan, Shandong
  - Yunnan Cancer Hospital, Kunming, Yunan

IPD SHARING:
Plan to Share IPD: Undecided